CLINICAL TRIAL: NCT03076606
Title: Nurses Ability to Assess Visual Acuity in Geriatric Consultation
Acronym: AVIGE
Status: Terminated | Type: Observational
Why Stopped: recruiting issues and unavailable ophtalmologists
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: AVIGE 16-114
Record Dates: First submitted 2017-03-06; First posted 2017-03-10 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2020-01

CONDITIONS: Visual Acuity; Accidental Fall; Aging; Nurse's Role

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ophthalmologist examination — ophthalmologist examination after geriatric consultation

SUMMARY:
Nurses participate to geriatric evaluations for falling patients. For these patients, it is recommended to evaluate,especially, visual acuity but this is not currently done because it is difficult to systematically combine with an ophthalmologic consultation.

The HAS french recommendations propose to detect visual acuity deficiency using Monoyer and Parinaud scales, without specifying the professional qualification. According to the nurse competence decree of State Graduates, "sensory disorders" screening is a "non-vulnerable" examination, and can be performed by nurses. Therefore, they can use these scales, after training.

We propose to evaluate the correlation between visual acuity scores obtained by nurses in geriatric consultations and an ophthalmologist.

This study should include 204 patients over 65 years, who have fallen at least twice in the last 12 months. These patients will benefit from an evaluation by an ophthalmologist, after the geriatric consultation.

ELIGIBILITY:
Inclusion Criteria:

* at least 2 falls in the last 12 months,
* applied in geriatric evaluation
* talking French
* affiliated to the social security system

Exclusion Criteria:

* not communicating
* illiterate
* Total blindness

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged 65 and over referred for Visual Acuity evaluation
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2020-05-04 (Actual); Study Completion 2020-05-04 (Actual)

PRIMARY OUTCOMES:
visual acuity values concordance between nurses and ophthalmologist | day 1
  On 2 (near and far) binocular values per patient with their usual glasses. Concordance is assessed on the assignment of patients to one of the 3 groups: ≤ 5 / 10e, 6-7 / 10 e, ≥ 8/10 e

SECONDARY OUTCOMES:
new diagnosis or ophthalmologic pathology aggravation | day 1
  Percentage of patients in whom new diagnosis or ophthalmologic pathology aggravation was identified
cognitive influence | day 1
  Compare the binocular visual acuity values agreement in each subgroup: with MMSE <18/30 and with MMSE ≥18/30

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No